CLINICAL TRIAL: NCT01159197
Title: Cognitive-Behavioral Therapy for Sleep Disturbance in Patients Undergoing Hemodialysis and Its Impacts on Their Inflammatory Cytokines, Oxidative Stress and Autonomic Dysfunction
Brief Title: Cognitive-Behavioral Therapy for Sleep Disturbance in Patients Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-97-D-093
Record Dates: First submitted 2010-05-24; First posted 2010-07-09 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2008-11

CONDITIONS: Insomnia; Depression; Inflammation
Keywords: sleep disturbance; cognitive behavioral therapy; inflammation; oxidative stress; hemodialysis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Inflammation; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cognitive behaviorial therapy (Experimental)
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — Participants who randomized into the CBT group will receive 18 30-minute tri-weekly treatment sessions of CBT during the 6-week period
  Other Names: cognitive behavioral therpy

SUMMARY:
Background

More than 50% of dialysis patients experience sleep disturbances that significantly affect quality of life, overall morbidity, and mortality. There is no effective therapy except hypnotics, which have notable side effects. Cognitive-behavioral therapy (CBT) is effective for treating peritoneal dialysis (PD) patients, the elderly and cancer patients with chronic insomnia, but its effectiveness has never been reported in hemodialysis (HD) patients and its impacts on the inflammatory cytokines, oxidative stress and autonomic dysfunction in this population are unknown. The investigators investigated the effectiveness of CBT in HD patients by assessing changes in sleep quality, inflammatory cytokines, oxidative stress and autonomic dysfunction.

Objects

This study is designed to assess the effectiveness of CBT on sleep disturbance in insomnias HD patients. The investigators also evaluate the impacts of CBT on the inflammatory cytokines, oxidative stress and autonomic dysfunction in these insomnias HD patients.

Methods

The investigators expected to recruit 80 insomnias HD patients undergoing maintenance HD for more than 3 months for the investigation. Besides, 40 HD patients without sleep disturbance will be recruited for comparison. Patients with sleep disturbance (N=80) was randomized to either intervention (CBT) group (N=40) or control group (N=40). Participants in CBT group will receive 6-week CBT while in control group and patients without sleep disturbance only receive sleep hygiene education. The subjects were assessed at baseline and after the intervention with the Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), Beck depression index (BDI) and the International Index of Erectile Function (IIEF) for men and the Index of Female Sexual Function (IFSF) for women; and inflammatory cytokines (serum IL-1β, IL-18, and TNF-α levels), oxidative stress (TBARS, Total antioxidant status and serum 8-OHdG) and autonomic dysfunction (Baroreflex sensitivity, BRS) were measured.

Expected results

The investigators expect that CBT can improve the sleep disturbance in HD patients and may change the inflammatory cytokines, oxidative stress and autonomic dysfunction after the intervention in insomnias HD patients.

DETAILED DESCRIPTION:
Sleep disturbance is common in patients with renal disease. According to previous studies, it occurs in more than 50% of chronic kidney disease (CKD) patients and those undergoing dialysis. 1, 2 Insomnia, restless legs syndrome (RLS), daytime sleepiness, and sleep apnea syndrome are common complaints; such sleep disturbances significantly affect the quality of life, overall morbidity, hospitalization, and mortality. 3-5 The main remedy for sleep disturbances, hypnotics, have notable side effects such as daytime sleepiness, psychological dependence, and drug-to-drug interactions, which make these drugs less than an optimal therapy. 6 Cognitive-behavioral therapy (CBT), the most widely used psychological intervention for insomnia, combines cognitive strategies such as stimulus control and relaxation training and has been proven to be effective for chronic insomnia in the elderly, cancer patients, and chronic pain sufferers7, 8. In most published articles CBT has been reported be superior to pharmacological and other behavioral therapies.9 In our previous investigation10, we found that the CBT was effective in PD patients with sleep disturbance presented with declined of Pittsburgh Sleep Quality Index (PSQI) and Fatigue Severity Scale (FSS); furthermore, the inflammatory cytokines, such as IL-1β, IL-18, TNF-α also declined after CBT in those insomnias PD patients. In previous studies, changes in cytokine release correlated with insomnia in patients undergoing hemodialysis11 or with breast cancer.12 Nevertheless, the effectiveness of CBT of sleep disturbance in insomnias HD patients is still not known.

In this study, we investigated the effectiveness of CBT for treatment of HD patients with insomnia by assessing changes in sleep quality subjectively through self-report questionnaires. The purpose of this study was to identify new therapeutic options for sleep disorders beyond hypnotics in HD patients. Because the association of sleep disturbance, oxidative stress and autonomic dysfunction in general population and patient with sleep apnea were demonstrated in previous investigations, we also investigate the possible impacts of CBT on the oxidative stress, autonomic dysfunction in these patients.

This study is designed to:

1. To evaluate the effectiveness of CBT for sleep disturbance in maintenance HD patients.
2. To evaluate the possible impacts of CBT on inflammatory cytokines, oxidative stress and autonomic dysfunction in insomnias HD patients. .
3. To compare the systemic inflammation, oxidative stress and autonomic dysfunction in HD patients with and without sleep disturbance.

Study designs and methods Eighty ESRD patients undergoing maintenance hemodialysis (HD) for more than 6 months with subjective complaint of sleep disturbance and screening PSQI ≥ 5 will be recruited for the investigation. Besides, 40 ESRD patients undergoing HD for more than 6 months without sleep disturbance will also be recruited as the population-base control group. Insomnias HD patients (N=80) will be randomized into interventional group (CBT group) and control group in 1:1 ratio in the following 6-week trial.

All participants (N=120) will receive questionnaires including Pittsburgh Sleep Quality Index (PSQI), Fatigue Severity Scale (FSS), Beck depression index (BDI) and the International Index of Erectile Function (IIEF) for men and the Index of Female Sexual Function (IFSF) and check-ups of baroreflex sensitivity (BRS) for autonomic dysfunction before the trial. Also, all of them will get fasting blood sampling at the initiation of trial in the morning before mid-week HD section for analysis of inflammatory cytokines (serum IL-1β, IL-18, and TNF-α levels) and oxidative stress (TBARS, Total antioxidant status and serum 8-OHdG). Participants with sleep disturbance will be randomized into CBT group and control group in 1:1 ratio and all of them receive sleep hygiene education before the trial. Participants who randomized into the CBT group will receive 6 1-hour weekly treatment sessions of CBT during the 6-week period. Participants who received hypnotics chronically before being recruited were maintained at the same dose of hypnotics during the therapy. After the 6-week trail, all participants will receive PSQI, FSS, BDI, IIEF, IFSF and BRS again and 2nd blood sampling for analysis of inflammatory cytokine and oxidative stress again. All the questionnaires, BRS and analyses of inflammatory cytokine and oxidative stress will be performed again 3 months after the trial for the long-term follow-up analysis. The details of investigation are demonstrated in Figure 1.

ELIGIBILITY:
Inclusion Criteria:

* under maintenance hemodialysis for more than 6 months
* subjective sleep complaints and screening PSQI ≥ 5

Exclusion Criteria:

* active medical condition (hospitalization/surgery)
* active malignancy
* active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
improvement of sleep disturbance/depression/anxiety | 6 weeks

SECONDARY OUTCOMES:
Changes of inflammatory cytokines/oxidative stress | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yuan Chen, M.D, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan, Taiwan